CLINICAL TRIAL: NCT03916497
Title: Quantification de l'immunité T Anti-CMV à l'Aide d'un Test IGRA Chez Des Patients greffés rénaux et Des Patients dialysés, Comparaison Avec Une Population de témoins
Brief Title: Anti-CMV Cellular Immunity Quantification Using an IGRA Test in Kidney Transplant récipients and Hemodialysis Patients, Comparison to Control Patients
Acronym: Quantiferon
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC19.002; 2019-A00101-56 (Other: ID RCB)
Record Dates: First submitted 2019-03-18; First posted 2019-04-16 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Quantiferon-CMV; Cytomegalovirus Infections; Kidney Transplant Infection; Hemodialysis
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1 : kidney transplant recipients (KTR)
  Interventions: Diagnostic Test: Quantiferon CMV
- Group 2 : hemodialysis patients
  Interventions: Diagnostic Test: Quantiferon CMV
- Group 3 : Control patients
  Interventions: Diagnostic Test: Quantiferon CMV

INTERVENTIONS:
Diagnostic Test: Quantiferon CMV — Evaluate and compare interferon gamma (IFNy) production by T CD8 cells exposed to CMV antigens in CMV seropositive kidney transplant recipients, hemodialysis and control patients

SUMMARY:
Evaluation of anti-CMV T cellular immunity using an IGRA test (Quantiferon-CMV test) in kidney transplant recipients and hemodialysis patients, comparison to control patients.

DETAILED DESCRIPTION:
Cytomegalovirus (CMV) infection is a common opportunistic complication after kidney transplantation (KT). It has been associated with high morbidity and mortality in kidney transplant recipients (KTR). Its actual management is only based on the humoral immunity : the main risk factor for CMV infection after KT is the association of a seropositive donor and a seronegative recipient (so-called "D+/R- mismatch").

However several studies have highlighted the essential role of cellular immunity to control CMV infection. The Quantiferon-CMV (QF-CMV) is an IGRA test (Interferon Gamma Releasing Assay) which evaluates T CD8 lymphocytes production of Interferon Gamma (IFNy) exposed to CMV antigens. Some studies have shown the possible interest of the QF-CMV in predicting CMV infection after antiviral prophylaxis discontinuation or when CMV viremia is detected.

However some limits have been underlined. First its positivity threshold hasn't been approved in KTR. Hemodialysis patients (HP) called to receive a renal allograft also suffered from altered immunity. No study has directly compared the QF-CMV value in KTR, HP and control patients.

That's why we propose evaluating the expression of basal cellular immunity against CMV (far from any active infection) in KTR and HP using the QF-CMV and comparing it to control patients population (not suffering from kidney dysfunction or immunosuppression).

ELIGIBILITY:
Inclusion Criteria :

* For all patients :

  * to be seropositive for CMV
  * to not be opposed to the study
* For kidney transplant recipients :

  * to have received a kidney graft for over 1 year
  * to have received an induction therapy at transplantation time by anti-lymphocytes antibodies and steroids
  * to be currently receiving immunosuppressive therapy by calcineurins inhibitors (tacrolimus or cyclosporine), mycophenolic acid with or without steroids
  * to not suffer from another cause of immunosuppression
* For hemodialysis patients :

  * to be treated by hemodialysis for end stage renal disease
  * without prior solid organ transplant history
  * to not suffer from another cause of immunosuppression
* For control patients :

  * with normal kidney function (estimated GFR > 90 ml/min)
  * to not suffer from another cause of immunosuppression

Exclusion Criteria :

* patient under guardianship or deprived of his liberty

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Kidney transplant recipients will be recruited among KTR followed in the Kidney transplant department of Grenoble University Hospital.
  Hemodialysis patients will be recruited among hemodialysis patients on the waiting list for a kidney transplant in the Kidney transplant department of Grenoble University Hospital.
  Control patients will be recruited among non-hemodialysis and non-kidney transplanted patients followed in the Grenoble University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Quantification of anti-CMV T cellular immunity in kidney transplant recipients, hemodialysis patients and control patients. | Single measurement at Day 0 of patient inclusion
  Quantification of IFNy level producted by T cells exposed to CMV antigens using a Quantiferon-CMV test in kidney transplant recipients, hemodialysis patients and control patients.

SECONDARY OUTCOMES:
Quantification of patient cellular immunity. | Single measurement at Day 0 of patient inclusion
  Quantification of lymphocytes subpopulations.
Evaluation of kidney transplant recipient exposure to immunosuppressive therapy. | Single collection at Day 0 of patient inclusion
  Assessment of last tacrolimus trough concentration.
Estimation of renal function. | Single measurement at Day 0 of patient inclusion
  Evaluation of estimated glomerular filtration rate by plasmatic creatinin dosage using CKD-EPI estimate.
Assessment of CMV donor humoral immunity in kidney transplant recipients. | Single collection at Day 0 of patient inclusion
  Assessment of donor CMV serology.

CONTACTS AND LOCATIONS:
Overall Officials: Lionel Rostaing, Principal Investigator — Centre Hospitalier Universitaire Grenoble-Alpes
Locations (1):
- Chu Grenoble Alpes, Grenoble, France

REFERENCES:
- [Background] Radha R, Jordan S, Puliyanda D, Bunnapradist S, Petrosyan A, Amet N, Toyoda M. Cellular immune responses to cytomegalovirus in renal transplant recipients. Am J Transplant. 2005 Jan;5(1):110-7. doi: 10.1111/j.1600-6143.2003.00647.x. PMID 15636618
- [Background] Lisboa LF, Kumar D, Wilson LE, Humar A. Clinical utility of cytomegalovirus cell-mediated immunity in transplant recipients with cytomegalovirus viremia. Transplantation. 2012 Jan 27;93(2):195-200. doi: 10.1097/TP.0b013e31823c1cd4. PMID 22179399
- [Background] Kumar D, Chernenko S, Moussa G, Cobos I, Manuel O, Preiksaitis J, Venkataraman S, Humar A. Cell-mediated immunity to predict cytomegalovirus disease in high-risk solid organ transplant recipients. Am J Transplant. 2009 May;9(5):1214-22. doi: 10.1111/j.1600-6143.2009.02618.x. PMID 19422346
- [Background] Manuel O, Husain S, Kumar D, Zayas C, Mawhorter S, Levi ME, Kalpoe J, Lisboa L, Ely L, Kaul DR, Schwartz BS, Morris MI, Ison MG, Yen-Lieberman B, Sebastian A, Assi M, Humar A. Assessment of cytomegalovirus-specific cell-mediated immunity for the prediction of cytomegalovirus disease in high-risk solid-organ transplant recipients: a multicenter cohort study. Clin Infect Dis. 2013 Mar;56(6):817-24. doi: 10.1093/cid/cis993. Epub 2012 Nov 29. PMID 23196955
- [Background] Cantisan S, Lara R, Montejo M, Redel J, Rodriguez-Benot A, Gutierrez-Aroca J, Gonzalez-Padilla M, Bueno L, Rivero A, Solana R, Torre-Cisneros J. Pretransplant interferon-gamma secretion by CMV-specific CD8+ T cells informs the risk of CMV replication after transplantation. Am J Transplant. 2013 Mar;13(3):738-45. doi: 10.1111/ajt.12049. Epub 2013 Jan 11. PMID 23311355
- [Background] Walker S, Fazou C, Crough T, Holdsworth R, Kiely P, Veale M, Bell S, Gailbraith A, McNeil K, Jones S, Khanna R. Ex vivo monitoring of human cytomegalovirus-specific CD8+ T-cell responses using QuantiFERON-CMV. Transpl Infect Dis. 2007 Jun;9(2):165-70. doi: 10.1111/j.1399-3062.2006.00199.x. PMID 17462006